CLINICAL TRIAL: NCT00497172
Title: An Italian Multicenter, Randomized, Single Blind Study of the Sirolimus Eluting Stent in the Treatment Of Diabetic Patients With De Novo Coronary Artery Lesions
Brief Title: Diabetes Drug Eluting Sirolimus Stent Experience in Restenosis Trial
Acronym: DESSERT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRDIT 00-02/02
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): drug-eluting stent
  Interventions: Device: CYPHER Sirolimus-eluting stent
- 2 (Active Comparator): bare-metal stent
  Interventions: Device: Bx SONIC bare metal stent

INTERVENTIONS:
Device: CYPHER Sirolimus-eluting stent — drug-eluting stent
  Arms: 1
Device: Bx SONIC bare metal stent — bare-metal stent
  Arms: 2

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the Sirolimus-eluting stent CYPHERTM and/or updated version in reducing angiographic in-stent late loss in de novo native coronary lesions of diabetic patients as compared to the bare metal Bx SONIC balloon-expandable stent.

The secondary objective is to assess cost-effectiveness expressed in incremental cost/life year gained or cost/quality adjusted life year gained at different time points (8 months, 1 year).

DETAILED DESCRIPTION:
This is a multicenter (11 centers), prospective, randomized single blind study. This study has a 2-arm design assessing the safety and effectiveness of the Sirolimus-eluting stent CYPHERTM and/or updated version to the bare metal Bx SONICTM stent. A total of 250 patients will be entered in the study and will be randomized on a 1:1 basis. Patients who meet the eligibility criteria will be either randomized to the Sirolimus-eluting stent or the bare metal Bx SONIC stent. The investigator cannot be blind because the outer appearance of the system for the implant of the Sirolimus-eluting stent differs from that of the bare metal stent and will therefore immediately be recognized by the surgeon. However the patient will not know which stent will be implanted. Patients will be followed at 30 days, 9 and 12 months post-procedure, with all patients undergoing repeat angiography at 8 months. Additionally, medical costs associated with the index hospitalization and length of stay, and repeat hospitalizations and costs associated with other relevant medical resource use during the 1 year follow-up period will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥ 18 years of age;
2. Female of childbearing potential must have a negative pregnancy test within 7days of enrollment and utilize reliable birth control for eight months after enrollment;
3. Patients with IDDM (Type I) treated for at least 3 months with documented HbA1c, or NIDDM (Type II) treated with oral antidiabetics for at least 3 months;
4. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia OR patient with previous (>24 hours) myocardial infarction with documented residual ischemia and/or viable myocardium;
5. Single or double stent treatment of de novo lesion in a major coronary artery in patients with single or multi-vessel disease; patients with multi-vessel disease can be included only if a maximum of two vessels require treatment with a maximum of three lesions in total, no more than two lesions per vessels. The two lesions in a single vessel must be >10 mm apart (visual estimate) and must be treated with the assigned stent.
6. Target vessel diameter at the lesion site is ≥ 2.50mm and ≤ 3.5mm in diameter (visual estimate);
7. Target lesion is ≥ 13mm and ≤ 25mm in length (visual estimate);
8. Target lesion stenosis is >50% and <100% (visual estimate);
9. At least TIMI II coronary flow;
10. Acceptable candidate for coronary artery bypass surgery (CABG);
11. Patient is willing to comply with the specified follow-up evaluation;
12. Patient must provide written informed consent prior to the procedure using a form that is approved by the local Ethics Committee;
13. Patient can be pretreated with aspirin and clopidogrel or, alternatively, aspirin alone plus a loading dose of 300 mg of clopidogrel before procedure completion in case of urgent PCI, and GPIIb IIIa inhibitors (Tirofiban or Abciximab)

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
2. Unprotected left main coronary disease with ≥50% stenosis;
3. Significant (>50%) stenoses proximal or distal to the target lesion that might require revascularization or impede runoff;
4. Have a target lesion in an arterial or venous by-pass graft;
5. Calcified lesion which cannot be successfully predilated;
6. Documented left ventricular ejection fraction ≤ 30%;
7. TIMI 0-I coronary flow ;
8. Impaired renal function (creatinine > 3.0 mg/dl) at the time of treatment;
9. Pretreatment with devices other than balloon angioplasty;
10. Target lesion has excessive tortuousity or angulation (>45°) which makes it unsuitable for stent delivery and deployment;
11. Target lesion involves bifurcation including a diseased side branch ≥2 mm in diameter (either stenosis of both main vessel and major branch or stenosis of just major branch) that would require side branch stenting;
12. Prior stent within 5mm of target lesion;
13. Direct Stenting;
14. Recipient of heart transplant;
15. Patient with a life expectancy less than 12 months;
16. Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix), heparin and GPIIb IIIa inhibitors (Tirofiban or Abciximab) stainless steel, contrast agent (that cannot be managed medically), or sirolimus;
17. Recent (6 months) cerebrovascular accidents or intracranial hemorrhage;
18. Any significant medical condition which in the investigator.s opinion may interfere with the patient.s optimal participation in the study;
19. Currently participating in an investigational drug or another device study;
20. Intervention of another lesion has occurred within 6 months before the index procedure;
21. In the investigator.s opinion, the lesion is not suitable for stenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-01; Primary Completion 2006-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
in-stent LL | 8-month post-procedure

SECONDARY OUTCOMES:
MACE | 1, 9, and 12 Months
Target vessel failure | 12 months
Target lesion or target vessel revascularization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: A. Maresta, MD, Principal Investigator — Azienda USL Ravenna
Locations (1):
- Azienda USL Ravenna - Ospedale santa Maria delle Croci, Ravenna, Italy